CLINICAL TRIAL: NCT04036097
Title: Prospective Stratification of Infectious Risks in Multiple Sclerosis (InRIMS-Study)
Brief Title: Prospective Stratification of Infectious Risks in Multiple Sclerosis
Acronym: InRIMS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Multiple Sclerosis Society (Unknown); Bangerter-Rhyner Stiftung (Unknown); Center for Chronic Immunodeficiency (CCI) in Freiburg, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-00465; me18Decard
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: secondary immunodeficiencies; disease-modifying treatments (DMT); immunosuppressive therapy; serious infection; respiratory tract infections (RTI); urinary tract infections; infection diary; Swiss MS Cohort (SMSC); SUMMIT (Serially Unified Multicenter Multiple Sclerosis Investigation) studies
MeSH Terms: conditions — Multiple Sclerosis; Respiratory Tract Infections; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MS-adapted AWIS questionnaire (MS-AWIS) — The predefined questionnaire-based infection score of the Airway Infection Susceptibility (AWIS) study is predictive for the occurrence of respiratory tract infections (RTI). In addition several MS-specific items (e.g. bladder dysfunction and urinary tract infections) are included into the AWIS questionnaire (MS-AWIS).
Other: infection diary (MS-AWIS diary) — MS patients prospectively fill out monthly infection diaries for 24 months. Infection diaries will either be sent back (with pre-franked envelopes) or handed back to the InRIMS-study team during regular clinical visits (usually every 6 or 12 months).

SUMMARY:
This monocentric study is to identify factors that increase the susceptibility for infections and establish a questionnaire-based infection score that allows a prospective stratification for infectious risks in patients with multiple sclerosis (MS) (InRIMS-Study). The study will utilize a validated, MS-adapted questionnaire and infection diary from the Airway Infection Susceptibility (AWIS) study in a regularly followed, prospective cohort of MS patients. It is a nested project of the prospective observational Swiss MS Cohort (SMSC) and SUMMIT (Serially Unified Multicenter Multiple Sclerosis Investigation) studies.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) for the InRIMS-study and Swiss MS Cohort (SMSC) and/or Serially Unified Multicenter Multiple Sclerosis Investigation (SUMMIT) study

Exclusion Criteria:

* Not able to sufficiently understand the patient information and questionnaire (German language)
* MS Patients with long-term antibiotic prophylaxis
* MS Patients with known primary immunodeficiency, under chemotherapy due to any malignancy or HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients participating in the SMSC or SUMMIT study with or without DMT
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
AWIS RTI score | Baseline
  AWIS RTI score is based on the data collected with the MS-adapted AWIS (MS-AWIS) questionnaire; score varies between 0 (no RTI burden) and 50 (maximal RTI burden)
infection diary score | 24 months
  monthly diary RTI score, averaging ten RTI symptom categories with the coding "0" for "no infection reported", "1" for "reported infection with duration < 2 weeks", and "2" for "reported infection present with duration >2 weeks

SECONDARY OUTCOMES:
Comparison of infection scores between patients receiving Disease Modifying Therapies (DMTs) and those who do not receive DMTs | 24 months
  Comparison of infection scores between patients receiving DMTs and those who do not receive DMTs

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Décard, Dr. med, Principal Investigator — University Hospital Basel, Department of Neurology
Locations (1):
- University Hospital Basel, Department of Neurology, Basel, Switzerland